CLINICAL TRIAL: NCT02879292
Title: Post-operative Outcomes in the Pyloromyotomy Procedure Under Spinal Anesthesia: A Retrospective Study in 100 Cases
Brief Title: Post-operative Outcomes in the Pyloromyotomy Procedure Under Spinal Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Other Study IDs: BnaiZionMC-16-LG-010
Record Dates: First submitted 2016-08-18; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Postoperative Pain
Keywords: Pyloric stenosis spinal anesthesia postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Spinal anesthesia — Spinal Anesthesia

SUMMARY:
Infantile hypertrophic pyloric stenosis (HPS) is one of the most common gastrointestinal medical emergencies.This retrospective study will review the files of all infants with HPS, who were treated by open pyloromyotomy under spinal anesthesia in the Bnai Zion Medical Center between the years 2006 to 2015.

DETAILED DESCRIPTION:
Infantile hypertrophic pyloric stenosis (HPS) is one of the most common gastrointestinal medical emergencies that occur during the first 2 months of life.

Anesthetic induction and airway management of infants with HPS can be challenging because of the accumulation of significant volumes of gastric content, predisposing these patients to pulmonary aspiration during the induction of general anesthesia Despite the correction of systemic metabolic alkalosis, cerebrospinal fluid can remain alkalotic, and in this context hyperventilation and opioids may increase the risks of post-operative central apnea. All of the above anesthetics risks urged some anesthetists to alternatively use spinal anesthesia (SA) in infants undergoing pyloromyotomy.

This anesthetic technique proved to be both safe and efficient in infants undergoing pyloromyotomy, in addition to decreasing the mentioned risks associated with the other techniques.

This retrospective study will review the files of all infants with HPS, who were treated by open pyloromyotomy under SA in the Bnai Zion Medical Center between the years 2006 to 2015. It is designed to evaluate the postoperative full enteral feeding time, pain management and the incidence of post-operative apnea, the incidence of substantial vomiting episodes and other spinal anesthesia complications as secondary outcomes in infants undergoing pyloromyotomy under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Infants with Hypertrophic Pylorostenosis, treated by open pyloromyotomy under Spinal Anesthesia

Exclusion Criteria:

Infants with Hypertrophic Pylorostenosis,treated by open pyloromyotomy under General Anesthesia

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants with Hypertrophic Pylorostenosis, who were treated by open pyloromyotomy under Spinal Anesthesia in the Bnai-Zion Medical Center between the years 2006 to 2015.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measure in numerical scale | till 24 hours after surgery

SECONDARY OUTCOMES:
Vomiting measure in numbers | till 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: mira koch, M.A., Study Chair — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Yes